CLINICAL TRIAL: NCT06436625
Title: Outpatient Pulmonary Rehabilitation in Patients With Advanced Stage Non-small Cell Lung Cancer Receiving Immunotherapy: a Randomized Controlled Trial (OPAL-study)
Brief Title: Outpatient Pulmonary Rehabilitation in Non-small-cell Lung Cancer Receiving Immunotherapy
Acronym: OPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Landsteiner Institute for Lung Research and Pneumological Oncology (Other)
Collaborators: Klinik Pirawarth (Unknown); Therme Wien Med (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OPAL Version 3.0
Record Dates: First submitted 2024-05-17; First posted 2024-05-31 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatient Pulmonary Rehabilitation (Active Comparator): The intervention group will receive 6 weeks of outpatient pulmonary rehabilitation in one of the rehabilitation centers (Therme Wien Med, Klinik Pirawarth in Wien).
  Interventions: Other: outpatient pulmonary rehabilitation
- Control (No Intervention): The control group receives no pulmonary rehabilitation since this is standard of care.

INTERVENTIONS:
Other: outpatient pulmonary rehabilitation — Patients undergo six weeks of an outpatient rehabilitation program in one of the rehabilitation centers (Therme Wien Med, Klinik Pirawarth in Wien).
  Arms: Outpatient Pulmonary Rehabilitation

SUMMARY:
The aim of this prospective study is to evaluate the effects of an outpatient pulmonary rehabilitation program on the quality of life, performance and tumor growth of metastatic lung cancer patients receiving ongoing immunotherapy.

The main questions it aims to answer are:

The primary objective of the study is to assess the effects of outpatient pulmonary rehabilitation (OPR) on exercise capacity measured by difference in the 6-minute walking test (6MWT) in patients with advanced stage lung cancer receiving immunotherapy measured by difference in the 6-minute walking test (6MWT).

Secondary endpoints in this study include progression free survival (PFS) and the effect of OPR on long term exercise capacity measured by 6MWT (difference in 6MWT after week 15 and 24).

Researchers will compare two groups of patients: one group of patients receives 6 weeks of outpatient pulmonary rehabilitation (intervention group), while the other patient group serves as control since this is standard of care to evaluate the effects of outpatient pulmonary rehabilitation.

DETAILED DESCRIPTION:
The effect of an outpatient pulmonary rehabilitation program on the quality of life, performance and tumor growth of metastatic lung cancer patients receiving ongoing immunotherapy will be investigated. Comparable data on rehabilitation under ongoing immunotherapy are almost non-existent in a prospective setting.

In addition, all patients with metastatic lung cancer could benefit from the study results if the benefit of outpatient rehabilitation can be proven in this patient population.

Patients will be randomized into two treatment arms and will be allocated due to randomization process. Both arms will receive standard-of care oncologic therapy according to national and international guidelines. In addition, one arm will receive 6 weeks of a standardized OPR (intervention group).

Patients who were randomized into the intervention group will be referred to one of the rehabilitation centers (Therme Wien Med or Klinik Pirawarth in Vienna) regarding of patients choice. The OPR is performed identical at both rehabilitation centers and according to Austrian guidelines (consistency was reassured by both heads of institutes).

Before the intervention (T0-baseline, week 0) patients will perform a 6-minute walking test (6MWT) (primary endpoint) together with additional secondary objective measurements (see section secondary endpoints or graphical overview). A follow-up will be performed after completion of OPR (T1, week 6) and every 9 weeks thereafter for the first 52 weeks (T1, FUP-T2, FUP-T3, FUP-T4-T6). After 52 weeks (FUP-T≥7) the intervals for follow-up visits is determined by the treating physician.

The end of study is reached if patient shows tumor progression (according to RECIST 1.1 criteria) after FUP-T3 (week 24) or - if patients has experienced tumor progression before FUP-T3 - after FUP-T3 (week 24).

ELIGIBILITY:
Inclusion criteria

* Capable and willing to give signed informed consent, which includes compliance with the requirements
* Age ≥ 18 years at the time of screening
* Histological or cytological confirmed non-squamous non-small cell lung cancer
* Previously untreated patients with histologically or cytologically documented metastatic (Stage IV according to Version 9 on the IASLC Staging Manual in Thoracic oncology) or recurrent NSCLC
* World Health Organization (WHO)/ECOG PS of 0 or 1 at enrollment
* At least 1 lesion not previously irradiated that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by CT or MRI scan must be performed within 28 days prior to randomization.
* Stable disease (SD), partial response (PR) or complete response (CR) (according to RECIST 1.1) after four cycles of first line chemo-immunotherapy and planned maintenance therapy
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies in advanced or metastatic therapy setting except ongoing first line immunotherapy

Exclusion criteria

* Physical or cognitive condition or symptoms that contraindicate execution of physical exercise or participation in a clinical exercise-based trial
* Symptomatic brain metastases
* Bone metastases with risk of pathological fracture with exercise training as assessed by treating physician
* Contraindication for immunotherapy
* Existence of more than one primary tumor such as: mixed small cell and NSCLC histology; synchronous or metachronous tumors that could represent distinct primary tumors
* Evidence of other active cancer disease
* Any medical condition that might be worsened by exercise training including, but not restricted to severe congestive heart failure (NYHA III/IV), unstable angina pectoris, myocardial infarction or cardiac surgery 6 months prior to randomization
* Major surgical procedure (as defined by the investigator) within 28 days prior to randomization or planned during the next 56 days
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walking Test | Measured at baseline and 8 weeks afterwards
  The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity and will be measured at baseline and 8 weeks afterwards.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival is defined as the time from therapy until the date of progressive disease using RECIST 1.1 assessments, or date of death due to any cause, whichever occurs first.
Six Minute Walking Test (longterm) | Measured at week 15 and 24
  Effect of OPR on long term exercise capacity measured by 6MWT (difference in 6MWT after week 15 and 24)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Illini, Dr., Principal Investigator — Karl Landsteiner Institute of Lung Research and Pulmonary Oncology, Klinik Floridsdorf
Locations (1):
- Klinik Floridsdorf, Abteilung für Innere Medizin und Pneumologie, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No